CLINICAL TRIAL: NCT03170739
Title: Effects of Dexmedetomidine and Dopamine on Renal Function After Selective Major Surgery in Adult Patients
Brief Title: Effects of Dexmedetomidine and Dopamine on Renal Function After Major Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tao Zhang (Other)
Responsible Party: Sponsor-Investigator, Tao Zhang, Clinical Professor of Department of Anesthesiology, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DexR
Record Dates: First submitted 2017-05-17; First posted 2017-05-31 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Renal Function
Keywords: dexmedetomidine; dopamine; surgery
MeSH Terms: interventions — Dexmedetomidine; Dopamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dexmedetomidine (Experimental): Dexmedetomidine 0.5ug/kg iv follow by 0.2ug/kg/h ivpump at the beginning of surgery.
  Interventions: Drug: Dexmedetomidine
- Dopamine (Experimental): Dopamine 3ug/kg/min ivpump at the beginning of surgery.
  Interventions: Drug: Dopamine
- Dexmedetomidine+dopamine (Experimental): Dexmedetomidine 0.5ug/kg iv follow by 0.2ug/kg/h ivpump, combined with dopamine 3ug/kg/min ivpump at the beginning of surgery.
  Interventions: Drug: Dexmedetomidine; Drug: Dopamine
- Control group (No Intervention): No intervention

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine given during surgery.
  Arms: Dexmedetomidine; Dexmedetomidine+dopamine
Drug: Dopamine — Dopamine given during surgery.
  Arms: Dexmedetomidine+dopamine; Dopamine

SUMMARY:
Acute kidney injury (AKI) is associated with complications that may lead to multiorgan dysfunction and potentially to multi-organ failure after major surgery. Dexmedetomidine is a highly selective alpha(2)-adreno receptor agonist widely used during anesthesia. In animals, dexmedetomidine has shown protective effects in AKI after surgery. Dopamine (DA) is an organic chemical of the catecholamine and phenethylamine families that has been widely used to increased renal blood flow and urine output during surgery. However, the clinical effects of dexmedetomidine and dopamine on renal function are still controversial. The aim of this study is to investigate whether dexmedetomidine and dopamine have positive effects on renal function after selective major surgery.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is associated with complications that may lead to multiorgan dysfunction and potentially to multi-organ failure in critically ill patients. AKI accounts for 5-10% after general surgery to 45% after cardiac surgery during hospital stays and tends to be associated with increased length of hospital stay as well as increased morbidity and mortality. Even slight increases in postoperative serum creatinine concentrations have been associated with almost 5-fold increases in mortality. Dexmedetomidine is a potent and highly selective alpha(2)-adreno receptor agonist that has analgesic, sedative, anxiolytic, and sympatholytic effects. In animals, dexmedetomidine has shown protective effects in several models of ischemia-reperfusion, which is thought to be the principal mechanism of AKI in the context of surgery. Dopamine (DA) is an organic chemical of the catecholamine and phenethylamine families that has been widely used to increased renal blood flow and urine output. However, the clinical effects of dexmedetomidine and dopamine on renal function are still controversial. The aim of this study is to investigate whether dexmedetomidine and dopamine have positive effects on renal function after selective major surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing selective major surgery

Exclusion Criteria:

* Patients undergoing urologic surgery or neurosurgery
* Patients with preoperative renal disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative renal function | Change from baseline to the 5th day after surgery
  Serum Cr and Cys-c
Mortality | 30 days
Postoperative complications | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Sun Yat-sen University, Guangzhou, China

REFERENCES:
- [Background] Ji F, Li Z, Young JN, Yeranossian A, Liu H. Post-bypass dexmedetomidine use and postoperative acute kidney injury in patients undergoing cardiac surgery with cardiopulmonary bypass. PLoS One. 2013 Oct 10;8(10):e77446. doi: 10.1371/journal.pone.0077446. eCollection 2013. PMID 24130886